CLINICAL TRIAL: NCT00658892
Title: B7-DC Xab Plasma Therapy for the Treatment of Metastatic Melanoma. A Feasibility/Pilot Study
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593085; P30CA015083 (NIH); MC0677 (Other: Mayo Clinic Cancer Center); 06-006992 (Other: Mayo Clinic IRB); NCI-2009-01343 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2008-04-12; First posted 2008-04-15 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Flow Cytometry; Immunologic Techniques

INTERVENTIONS:
Biological: B7-DC cross-linking antibody rHIgM12B7
Other: flow cytometry
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This clinical trial is studying the side effects and best dose of a monoclonal antibody in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety/toxicity of a single dose of B7-dendritic cell cross-linking antibody containing plasma in treating patients with stage IV melanoma.

Secondary

* Describe the immunological changes (Th1/Th2 balance, frequency of tumor specific cytotoxic T lymphocytes, and plasma cytokine profiles) in the treated patients.
* Determine the treatment impact on tumor growth (e.g., objective response, time to progression).

OUTLINE: Patients receive B7-dendritic cell cross-linking antibody IV once on day 1.

Patients undergo peripheral blood collection at baseline and periodically after infusion for analysis of dendritic cell activation, cytotoxic T-lymphocyte activity, immune cell impact, and serum cytokine changes using immunophenotyping and flow cytometry.

After completion of study treatment patients are followed every 2 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Stage IV disease (M1a and M1b only)
* Measurable disease according to RECIST criteria
* HLA-A2 positive
* Must have IgA in serum (any concentration)
* No known standard therapy for this disease that is potentially curative or proven capable of extending life expectancy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin ≥ 10.0 g/dL
* Platelet count ≥ 75,000/mm^3
* AST ≤ 5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to provide informed consent
* Agrees to return to Mayo Clinic Rochester for follow-up
* Agrees to participate in the mandatory translational research component of the study
* No uncontrolled or current infection
* No known immune deficiency
* No B or AB blood grouping

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy and recovered
* More than 4 weeks since prior biologic therapy
* No concurrent immunosuppressive therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-04-08 (Actual); Primary Completion 2010-02-15 (Actual); Study Completion 2012-05-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of B7-dendritic cell cross-linking antibody

SECONDARY OUTCOMES:
Progression free survival and overall survival time
Toxicity
Tumor response in terms of complete or partial response at 8 weeks
Tetramer response
Percent change in the number of T, B, NK cells, monocytes and dendritic cells from pretreatment levels as well as the percent change in plasma concentrations of various molecular components

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States